CLINICAL TRIAL: NCT05591664
Title: Comparison of Eicosapentaenoic Acid Serum Levels in Patients With Gestational Diabetes and Control Group
Brief Title: Eicosapentaenoic Acid Serum Levels in Patients With Gestational Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Senol Senturk, Associate professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2022/170
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; Eikosapentaenoik acid; fatty acids; omega-3
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1: There will be 38 patients diagnosed with gestational diabetes in the study group.
  Interventions: Diagnostic Test: eicosapentaenoic acid
- GROUP 2: There will be 80 normal pregnant women in the control group
  Interventions: Diagnostic Test: eicosapentaenoic acid

INTERVENTIONS:
Diagnostic Test: eicosapentaenoic acid — eicosapentaenoic acid levels of the groups will be monitored

SUMMARY:
In this study, we aim to compare the blood levels of Eicosapentaenoic acid (EPA) in gestational diabetes patients with normal pregnant women, to reveal the relationship between these markers, which are known to be effective on metabolic function, and gestational diabetes, and to contribute to future studies and possible treatment options.

DETAILED DESCRIPTION:
The research is a prospective cross-sectional study to be conducted at Recep Tayyip Erdogan University Training and Research Hospital, Department of Obstetrics and Gynecology. The current treatments of the patients will not be changed and no medical treatment or interventional procedures will be applied to the patients for study purposes. After the patients are informed about the study, their signatures will be taken on the consent form stating that they voluntarily participated in the study. Apart from the biochemical parameters required for the diagnosis and treatment of the patients, different parameters will not be considered. The supply of Eicosapentaenoic acid (EPA) kits required for the study will be provided by the executive physician and the blood taken from the patients will be evaluated.

G * Power 3.1.9.7 program was used to calculate the sample size for this study. At 80% statistical power and α=0.05 significance level, the smallest required sample size was calculated as 110 (control :75- study :35) when d=0.51 effect size was calculated according to t-test for independent groups. Considering that there may be missing data, 118 women between the ages of 18-46 will be included in the study. There will be 38 patients diagnosed with gestational diabetes in the study group. There will be 80 normal pregnant women in the control group. The diagnosis of GDM cases will be determined by 75 g oral glucose tolerance test (OGTT) performed between 24 and 28 weeks of gestation. According to the International Association of Diabetes and Pregnancy Study Groups (IADPSG) criteria, pregnant women will be considered to have GDM if one of the following plasma glucose values is met or exceeded: 0.st ≥92 mg/dl; 1st hour ≥180 mg/dl; 2nd hour ≥153 mg/dl.

Demographic, clinical and laboratory data of the pregnant women included in the study, age, number of previous live-stillbirths, previou type of delivery, gestational weeks, complete blood count for each patient. Detailed anamnesis, including information such as family history of diabetes, will be recorded. The last menstrual period, obstetric examination and ultrasonography findings will be taken as basis in the determination of the gestational week.

Inclusion criteria of patients in the study: 18-46 years old pregnant women at 24-28. gestational weeks Exclusion criteria of the patients in the study: For each group; Pregnant women under 18-46 years of age, multiple pregnancies, stillbirth, presence of preeclampsia, pregestational diabetes mellitus, hypertension, history of congenital cardiopathy, presence of serious systemic disorders such as chronic liver and kidney diseases, active smoking, being a smoker will be determined.

Since the medical treatment of the patients was not changed and additional medical treatment and interventional procedures were not applied in the study, it would not be necessary to take safety precautions. The blood taken from the patients for routine diagnosis and treatment will be stored at -20 degrees Celsius after the serum and plasma are separated. By comparing the blood levels of Eicosapentaenoic acid (EPA) in gestational diabetes patients with normal pregnant women, the relationship between these markers, which are known to be effective on metabolic function, and gestational diabetes will be evaluated. Afterwards, follow-up, treatment and laboratory evaluation for study purposes are not required.

ELIGIBILITY:
Inclusion Criteria: 18-46 years old pregnant women at 24-28 weeks of gestation -

Exclusion Criteria: For each group; Pregnant women under 18 or over 46 years of age, multiple pregnancies, stillbirth, presence of preeclampsia, pregestational diabetes mellitus, hypertension, history of congenital cardiopathy, presence of serious systemic disorders such as chronic liver and kidney diseases, active smoking, being a smoker will be determined

-

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-46 years old pregnant women at 24-28 weeks of gestation with and without gestational mellitus (study and control)
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
eicosapentaenoic acid | 6 months
  eicosapentaenoic acid levels between groups will be measured

CONTACTS AND LOCATIONS:
Overall Officials: SENOL SENTURK, Study Director — Recep Tayyip Erdogan University

IPD SHARING:
Plan to Share IPD: Undecided